CLINICAL TRIAL: NCT06769789
Title: Evaluation of Pregnancy Outcome in Poor Responder Patients in IVF Cycle with Usage of Drug-free In-vitro Activation of Follicles Ovary
Brief Title: Evaluation of Pregnancy Outcome with Usage of Drug-free In-vitro Activation of Follicles Ovary
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malihe Mahmoudinia (Other)
Responsible Party: Sponsor-Investigator, Malihe Mahmoudinia, Associate Professor of obstetrics & Gynecology, Fellowship of infertility, Faculty of Medicine, Mashhad University of Medical Sciences, Mashhad, Iran, Mashhad University of Medical Sciences
Organization: Mashhad University of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.MUMS.IRH.REC.1403.127
Record Dates: First submitted 2024-12-22; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Infertility (IVF Patients); Infertile Females or Females with Ovarian Insufficiency
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Drug -free invitro activation of ovary in women (Experimental)
  Interventions: Other: Drug free invitro activation Ovary

INTERVENTIONS:
Other: Drug free invitro activation Ovary — Drug free invitro activation Ovary

SUMMARY:
This study is the pilot study to evaluate the effect of Drug-free in vitro activation to improve the outcomes of IVF in poor responder women

DETAILED DESCRIPTION:
First, patients who are poor responders based on Poseidon criteria 1, 3 (women under 35 years of age who either have abnormal ovarian reserve tests or have not had an adequate ovarian response in an IVF cycle) are included in the list of poor responders and are consulted after a complete evaluation by a physician. The patient has a history of poor response in previous IVF cycles. After obtaining the patient's consent, the patient undergoes laparoscopy. The laparoscopy procedure will be performed at Milad Infertility Center, which is equipped with a laparoscopy operating room and a laboratory nearby. The procedures will be performed by a single surgical team that includes laparoscopy and infertility flowsheets. After general anesthesia and pre- and post-operative care, double puncture laparoscopy will be performed. Two minor trocars will be placed, which will be held in place by an ovarian grasper. With scissors, a part of the ovarian cortex is first separated from the underlying medulla and strips of cortex 1 to 2 mm thick and 10 mm long are removed. They are immediately transferred to the adjacent laboratory. A 1 x 5 mm sample from the removed piece is used for histological examination and determination of the number of remaining follicles. The tissue is then divided into 1 x 1 x 1 mm pieces. The removal site will be sutured in case of bleeding. The preparation of the ovary into small pieces will be performed by a single physician for all patients. The prepared pieces are immediately transferred to the operating room. Then the surgeon places the prepared pieces in the tunnel between the cortex and medulla in the opposite ovary and then sutured. The patient is then followed up and immediately treated with FSH (Sinagene Company, Tehran, Iran) at a maximum dose of 300 units, and then the dose is adjusted according to the ovarian response. When a 12 mm follicle is observed, 0.25 mg of Sterotide (Merck Serono, Mississauga, Canada) is started. When the size of 1 or 2 follicles reaches 16, 10,000 units of HCG (Puyish Daru Company, Tehran, Iran) and two ampoules of Deca (Decapeptyl 0.2 mg, Ferring, Germany) are given together for triggering. Ovulation is performed 36 hours later under transvaginal ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* Women under 35 years of age who have one of the following characteristics:

Or poor response to gonadotropins in a previous IVF cycle (fewer than 3 oocytes in a previous IVF cycle)

Or ovarian reserve test AMH less than 1.1

Exclusion Criteria:

* Unwillingness to continue working with the researcher during the procedure

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 23 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
The number of oocytes obtained at oocyte pick-up (OPU) | Within 3 weeks after ovarian stimulation
Number of embryos | Within 3 weeks after ovarian stimulation
Quality of embryos at the end of IVF treatment | Within 3 weeks after ovarian stimulation
  A grade embryo was defined to have four blastomeres on the second day and seven or eight blastomeres on the third day with equal size and <20% fragmentation (high quality). Blastocyst embryos were assessed according to Gardner's criteria.

SECONDARY OUTCOMES:
Implantation rate | 4-8 weeks after transfer
Clinical pregnancy rate | one month after transfer
Miscarriage rate | 20 weeks after transfer

IPD SHARING:
Plan to Share IPD: No